CLINICAL TRIAL: NCT07269106
Title: Efficacy and Safety of Anrikefon for Postoperative Analgesia in Ophthalmic Surgery: A Multicenter, Randomized, Parallel-Control, Non-Inferiority Trial
Brief Title: Efficacy and Safety of Anrikefon for Postoperative Analgesia in Ophthalmic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiaoliang Gan, Director of the Department of Anesthesiology, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT2025115
Record Dates: First submitted 2025-11-17; First posted 2025-12-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Ophthalmic Surgery; Postoperative Pain Management; Opioid Analgesia
MeSH Terms: interventions — Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Anrikefon Group (Experimental): Intravenous injection of Anrikefon 1 μg/kg will be administered 15 minutes before the end of surgery
  Interventions: Drug: Anrikefon
- The Nalbuphine Group (Active Comparator): Intravenous injection of nalbuphine 0.1 mg/kg will be administered 15 minutes before the end of surgery
  Interventions: Drug: Nalbuphine

INTERVENTIONS:
Drug: Anrikefon — Anrikefon is a novel peripherally KOR agonist independently developed in China. In this study, anrikefon will be administered intravenously at a dose of 1 μg/kg, 15 minutes before the end of surgery.
  Arms: The Anrikefon Group
Drug: Nalbuphine — Nalbuphine is a traditional central KOR agonist with mixed μ-opioid receptor antagonist activity. In this study, nalbuphine will be administered intravenously at a dose of 0.1 mg/kg, 15 minutes before the end of surgery.
  Arms: The Nalbuphine Group

SUMMARY:
The goal of this clinical trial is to learn if Anrikefon works as well as nalbuphine to control postoperative pain in adults undergoing ophthalmic surgery under general anesthesia. It will also learn about the safety and recovery outcomes of using Anrikefon.

The main questions it aims to answer are:

* Does Anrikefon provide pain relief that is not inferior to nalbuphine after ophthalmic surgery?
* Does Anrikefon cause fewer central side effects, such as sedation or dizziness, compared with nalbuphine?
* Does Anrikefon help patients recover and get discharged faster after day-surgery procedures? Researchers will compare Anrikefon to nalbuphine to see if Anrikefon can offer effective and safer perioperative analgesia for ophthalmic day-surgery patients.

Participants will:

* Receive either an intravenous dose of Anrikefon or nalbuphine during surgery.
* Be monitored for pain scores, side effects, and recovery parameters after surgery.
* Complete follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for ophthalmic surgery under general anesthesia.
* Aged 18 to 70 years.
* With American Society of Anesthesiologists (ASA) physical status I to III.
* Body mass index (BMI) between 18 and 30 kg/m²
* Agree to participate in the trial and provide written informed consent.

Exclusion Criteria:

* History of cardiovascular or cerebrovascular events within the past 6 months, including unstable angina, ischemic myocardial infarction, or heart failure; or current presence of uncontrolled hypertension (>180/110 mmHg), aneurysm, or severe cardiac arrhythmia.
* Severe respiratory diseases such as pulmonary fibrosis, severe pulmonary abscess, cor pulmonale, or advanced chronic obstructive pulmonary disease (COPD).
* Significant neurological disorders such as brain injury or seizures, as well as severe psychiatric illnesses.
* Known allergy to kappa opioid receptor agonists or to general anesthetic agents used in this study.
* Current peptic ulcer disease, gastrointestinal bleeding, or known hypersensitivity to nonsteroidal anti-inflammatory drugs (NSAIDs), such as flurbiprofen axetil or paracetamol.
* Prior use of opioid or non-opioid analgesics, with the last administration occurring within five half-life periods of the drug.
* Continuous use of opioid analgesics for more than 10 days within the 3 months prior to screening.
* Use of drugs with unknown half-life periods that may affect analgesic efficacy within 14 days before randomization.
* History of major surgery within the past 3 months that may interfere with postoperative pain assessment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2026-01-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative pain severity at rest during the first 6 hours after surgery, measured with the Numeric Rating Scale (0-10, higher scores = worse pain) | In the PACU and at 1 , 2 , 4 and 6 hours after surgery
  Pain intensity at rest is recorded with the Numeric Rating Scale (NRS: 0 = no pain, 10 = worst possible pain). The area under the curve (AUC) for these scores will be calculated with the trapezoidal rule, using assessments performed in the PACU and at 1 , 2 , 4 and 6 hours post-operatively. A higher AUC indicates greater cumulative pain over the 6-hour period.

SECONDARY OUTCOMES:
Pain severity at rest and during eye movement, measured with the Numeric Rating Scale (0-10, higher scores = worse pain) | In the PACU and at 1, 2, 4, 6, 12 and 24 hours, as well as 1 week and 1 month postoperatively
  Participants rate their pain intensity at rest and again during voluntary eye movement using the Numeric Rating Scale (NRS: 0 = no pain, 10 = worst possible pain). Assessments are performed in the PACU and at 1, 2, 4, 6, 12, 24 hours, 1 week, and 1 month post-operatively. Higher scores indicate greater pain.
Cumulative pain severity during eye movement (0-6 hours) and at rest/during eye movement (0-12 hours and 0-24 hours), measured with the Numeric Rating Scale | In the PACU and at 1, 2, 4, 6, 12, and 24 hours postoperatively
  The area under the curve (AUC) is computed with the trapezoidal rule, multiplying the average Numeric Rating Scale within each interval by its duration and summing the products; a higher AUC indicates greater cumulative pain.
Cumulative consumption of rescue analgesics (flurbiprofen axetil in the PACU and paracetamol after discharge from the PACU) within 6, 12, and 24 hours postoperatively, as well as the time to first use | At 6, 12, and 24 hours postoperatively
  In-hospital, participants with resting NRS ≥4 will receive intravenous flurbiprofen axetil 1 mg/kg. Additional doses can be given if ≥3 hours have passed since the previous flurbiprofen dose and ≥1 hour since the last study drug. Breakthrough pain (NRS ≥7) may be treated immediately. Out-of-hospital, participants with resting NRS ≥4 will receive paracetamol 500 mg per dose, up to 2 g per day.
Percentage of patients not requiring rescue analgesics | At 6, 12, and 24 hours postoperatively
  During the 6-, 12-, and 24-hour postoperative periods, each patient's use of rescue analgesics (flurbiprofen axetil or paracetamol) is recorded. Patients not receiving rescue analgesics are classified as 'not used,' and the percentage is calculated for each group to evaluate postoperative analgesia adequacy.
Satisfaction score of analgesia within 24 hours postoperatively | Within 24 hours postoperatively
  A trained study assistant assessed satisfaction score of analgesia at rest using a 0 to 10 NRS scale, where 0 indicates 'completely dissatisfied' and 10 indicates 'completely satisfied.'
Emergence time | Through surgery completion, an average of 1 hour.
  Emergence time is defined as the interval from stopping anesthetics to eye opening or following simple commands.
PACU stay time | Through surgery completion, an average of 2 hours.
  PACU stay time is defined as the duration from arrival in PACU to the time of a modified Aldrete score of 9 or 10.
Time to first ambulation | Through surgery completion, an average of 24 hours.
  Time to first ambulation is defined as the interval from the completion of surgery to the patient's first episode of spontaneous mobilization (i.e., getting out of bed and initiating independent movement).
Postoperative hospital stay | Through surgery completion, an average of 24 hours
  Postoperative hospital stay (or in-hospital stay for day-surgery patients) is defined as the interval from the completion of surgery to formal discharge from the hospital.
Incidence of postoperative complications in the PACU and within 24 hours postoperatively | In the PACU and within 24 hours postoperatively
  All assessments of adverse events and medication records will be conducted under double-blind conditions, with evaluators blinded to participant group assignment. The incidence of adverse events will be calculated based on the total number of enrolled participants in each group.
Postoperative 24-hour recovery quality assessed using the 15-item Quality of Recovery questionnaire (QoR-15) | At 24 hours postoperatively
  Postoperative recovery was assessed using the QoR-15 questionnaire.
Intraocular pressure (IOP) [mmHg] | At 24 hours, 1 week, and 1 month postoperatively
  Measured with non-contact tonometer; higher values indicate elevated IOP.
Orbital pressure [digital palpation grade] | At 24 hours, 1 week, and 1 month postoperatively
  Graded by single examiner via digital palpation.
Uncorrected visual acuity (UCVA) [LogMAR] | At 24 hours, 1 week, and 1 month postoperatively
  Assessed with standard LogMAR chart; lower LogMAR indicates better acuity.
Best-corrected visual acuity (BCVA) [LogMAR] | At 24 hours, 1 week, and 1 month postoperatively
  Assessed with standard LogMAR chart after refraction; lower LogMAR indicates better acuity.

OTHER OUTCOMES:
Mechanical pain threshold of the operative eye at 2 and 24 hours postoperatively | At 2 and 24 hours postoperatively
  Quantitative assessment around the periocular area of the operative eye using electronic Von Frey test.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Zhongshan Ophthalmic Center, Sun Yat-Sen University, Guangzhou, Guangdong
  - The Affiliated Hospital of Yunnan University, Kunming, Yunnan
  - Eye & ENT Hospital of Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] An introductory note to the CHMP guidelines: choice of the non-inferiority margin and data monitoring committees by David Brown, Peter Volkers and Simon Day, Statistics in Medicine 2006; 25:1623-1627. Stat Med. 2007 Jan 15;26(1):230-3; author reply 234-5. doi: 10.1002/sim.2665. No abstract available. PMID 16900566
- [Result] Piaggio G, Elbourne DR, Pocock SJ, Evans SJ, Altman DG; CONSORT Group. Reporting of noninferiority and equivalence randomized trials: extension of the CONSORT 2010 statement. JAMA. 2012 Dec 26;308(24):2594-604. doi: 10.1001/jama.2012.87802. PMID 23268518
- [Result] Zhong Y, Xu Y, Lei Q, Yang M, Wang S, Hu X, Xie H, Li Y, Qin Z, Gu Z, Zhang J, Wang Y, Wu J, Wang H, Ming Y, Xia Z, Zhai H, Jiang K, Zhang P, Wang Z, Wang L, Li L, Cheng Z, Jiang H, Wang G, Chen J, Zhao Z, Chen X, Yan M. HSK21542 in patients with postoperative pain: two phase 3, multicentre, double-blind, randomized, controlled trials. Nat Commun. 2025 May 24;16(1):4830. doi: 10.1038/s41467-025-60013-y. PMID 40413233
- [Result] Wang X, Gou X, Yu X, Bai D, Tan B, Cao P, Qian M, Zheng X, Wang H, Tang P, Zhang C, Ye F, Ni J. Antinociceptive and Antipruritic Effects of HSK21542, a Peripherally-Restricted Kappa Opioid Receptor Agonist, in Animal Models of Pain and Itch. Front Pharmacol. 2021 Nov 16;12:773204. doi: 10.3389/fphar.2021.773204. eCollection 2021. PMID 34867403
- [Result] Shao R, Wang HY, Ruan ZR, Jiang B, Yang DD, Hu Y, Xu YC, Yang JT, Gao W, Zhao WY, Yan M, Lou H. Phase I clinical trial evaluating the safety, tolerance, pharmacokinetics and pharmacodynamics of HSK21542 injection in healthy volunteers. Basic Clin Pharmacol Toxicol. 2024 Dec;135(6):743-754. doi: 10.1111/bcpt.14094. Epub 2024 Oct 13. PMID 39397291
- [Result] Gou X, Chen Y, Ye Q, Meng Q, Jia Y, Li P, Wang Q, Wang J, Zhang C, Wang J, Dong Y. Preclinical evaluation of abuse potential of the peripherally-restricted kappa opioid receptor agonist HSK21542. Regul Toxicol Pharmacol. 2024 Dec;154:105731. doi: 10.1016/j.yrtph.2024.105731. Epub 2024 Oct 23. PMID 39455048
- [Result] Wang K, Chen M, Xu F, Zhang F, Liu L, Liu X, Sun Z, Zhao W, Wang Y, Yang J. Population pharmacokinetic modeling and exposure-response analysis of anrikefon: insights and implications in clinical analgesia. Expert Rev Clin Pharmacol. 2025 Jan-Feb;18(1-2):77-88. doi: 10.1080/17512433.2025.2449983. Epub 2025 Jan 23. PMID 39825476
- [Result] Zhang XM, Lun MH, Du W, Ma F, Huang ZQ. The kappa-Opioid Receptor Agonist U50488H Ameliorates Neuropathic Pain Through the Ca2+/CaMKII/CREB Pathway in Rats. J Inflamm Res. 2022 May 23;15:3039-3051. doi: 10.2147/JIR.S327234. eCollection 2022. PMID 35645576
- [Result] Li J, Ye H, Shen W, Chen Q, Lin Y, Gan X. Retrospective analysis of risk factors of postoperative nausea and vomiting in patients undergoing ambulatory strabismus surgery via general anaesthesia. Indian J Anaesth. 2020 May;64(5):375-382. doi: 10.4103/ija.IJA_16_20. Epub 2020 May 1. PMID 32724245
- [Result] Ye H, Lian X, Chen R, Zhu Y, Chen H, Huang J, Xie L, Ma W, Yang H, Guo W. Intraoperative administration of intravenous flurbiprofen axetil with nalbuphine reduces postoperative pain after orbital decompression: a single-center, prospective randomized controlled trial. J Pain Res. 2019 Feb 14;12:659-665. doi: 10.2147/JPR.S187020. eCollection 2019. PMID 30863138
- [Result] Ye Z, Zhu Y, Zhang R, Wang Y, Huang J, Gan X. Effect of Multimodal Preemptive Analgesia of Flurbiprofen Axetil, Nalbuphine, and Retrobulbar Block on Postoperative Pain and Enhanced Recovery in Patients Undergoing Oculoplastic Day Surgery: A Prospective, Randomized, Double-Blinded Study. Ophthalmic Plast Reconstr Surg. 2023 May-Jun 01;39(3):260-265. doi: 10.1097/IOP.0000000000002308. Epub 2023 Jan 24. PMID 36727809
- [Result] Charlson ES, Feng PW, Bui A, Grob S, Tao JP. Opioid Prescribing Patterns Among American Society of Ophthalmic Plastic and Reconstructive Surgery Members in the Medicare Part D Database. Ophthalmic Plast Reconstr Surg. 2019 Jul/Aug;35(4):360-364. doi: 10.1097/IOP.0000000000001266. PMID 30439721
- [Result] Shanthanna H, Ladha KS, Kehlet H, Joshi GP. Perioperative Opioid Administration. Anesthesiology. 2021 Apr 1;134(4):645-659. doi: 10.1097/ALN.0000000000003572. PMID 32991672
- [Result] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Result] Zhang L, Shu R, Zhao Q, Li Y, Wang C, Wang H, Yu Y, Wang G. Preoperative But Not Postoperative Flurbiprofen Axetil Alleviates Remifentanil-induced Hyperalgesia After Laparoscopic Gynecological Surgery: A Prospective, Randomized, Double-blinded, Trial. Clin J Pain. 2017 May;33(5):435-442. doi: 10.1097/AJP.0000000000000416. PMID 27518488
- [Result] Rohi A, Olofsson MET, Jakobsson JG. Ambulatory anesthesia and discharge: an update around guidelines and trends. Curr Opin Anaesthesiol. 2022 Dec 1;35(6):691-697. doi: 10.1097/ACO.0000000000001194. Epub 2022 Oct 3. PMID 36194149
- [Result] Raeder J. Procedure-specific and patient-specific pain management for ambulatory surgery with emphasis on the opioid crisis. Curr Opin Anaesthesiol. 2020 Dec;33(6):753-759. doi: 10.1097/ACO.0000000000000922. PMID 33027075
- [Result] Fan ZG, Zhang DD, Li ZW, Yang Y, Lin XF. Outpatient Surgery in Zhongshan Ophthalmic Center: Promise and Problems. Chin Med J (Engl). 2017 Jul 5;130(13):1623-1624. doi: 10.4103/0366-6999.208237. No abstract available. PMID 28639583
- [Result] Zhu Y, Li Z, Chen W, Fan P, Yang S, Liu X, Guo W, Gan X. Incidence and Risk Factors of Moderate to Severe Postoperative Pain Following the Placement of Primary and Secondary Orbital Implants: A Prospective Observational Study. Ophthalmic Plast Reconstr Surg. 2021 Jan-Feb 01;37(1):27-32. doi: 10.1097/IOP.0000000000001664. PMID 32282646
- [Result] Ye H, Chen R, Lian X, Huang J, Mao Y, Lu R, Ai S, Ma W, Lin J, Yang H, Guo W. Risk factors associated with postoperative pain and discomfort in oculoplastic surgery with general anesthesia: a prospective study. J Pain Res. 2018 Feb 21;11:407-415. doi: 10.2147/JPR.S156104. eCollection 2018. PMID 29503577
- [Result] Henzler D, Kramer R, Steinhorst UH, Piepenbrock S, Rossaint R, Kuhlen R. Factors independently associated with increased risk of pain development after ophthalmic surgery. Eur J Anaesthesiol. 2004 Feb;21(2):101-6. doi: 10.1017/s0265021504002042. PMID 14977340
- [Result] Lesin M, Sundov ZD, Jukic M, Puljak L. Postoperative pain in complex ophthalmic surgical procedures: comparing practice with guidelines. Pain Med. 2014 Jun;15(6):1036-42. doi: 10.1111/pme.12433. Epub 2014 Mar 25. PMID 24666698
- [Result] Fregoso G, Wang A, Tseng K, Wang J. Transition from Acute to Chronic Pain: Evaluating Risk for Chronic Postsurgical Pain. Pain Physician. 2019 Sep;22(5):479-488. PMID 31561647
- [Result] Tan Z, Dong Y, Li Q. Dynamics of Acute Postsurgical Pain over the Last Decade: A Bibliometric Analysis. Pain Res Manag. 2022 Nov 7;2022:8090209. doi: 10.1155/2022/8090209. eCollection 2022. PMID 36385903
- [Result] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004
- [Result] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Result] Weiser TG, Haynes AB, Molina G, Lipsitz SR, Esquivel MM, Uribe-Leitz T, Fu R, Azad T, Chao TE, Berry WR, Gawande AA. Estimate of the global volume of surgery in 2012: an assessment supporting improved health outcomes. Lancet. 2015 Apr 27;385 Suppl 2:S11. doi: 10.1016/S0140-6736(15)60806-6. Epub 2015 Apr 26. PMID 26313057